CLINICAL TRIAL: NCT04072263
Title: Adoptive T Cell Therapy in Patients With Recurrent Ovarian Cancer
Acronym: OVACURE
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, J.R. Kroep, MD PhD, Leiden University Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OVACURE
Record Dates: First submitted 2019-08-27; First posted 2019-08-28 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Ovarian Cancer Recurrent
MeSH Terms: interventions — Interferon alpha-2; Carboplatin; Paclitaxel

STUDY DESIGN:
Intervention Model Description: Carboplatin-paclitaxel day1, q3 weeks, 6x, plus TIL starting 14 days after the 2nd chemotherapy cycle, q3 weeks, 3x.
  Minus or plus:
  IFNα (3x10e6 U daily) starting one week before the first TIL infusion for 12 weeks in total.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): * Carboplatin-paclitaxel day1, q3 weeks, 6x, plus
  * Tumor Infiltrating Lymphocytes (TIL) starting 14 days after the 2nd chemotherapy cycle, q3 weeks, 3x.
  Interventions: Biological: Tumor Infiltrating Lymphocytes (TIL); Drug: Carboplatin; Drug: Paclitaxel
- Cohort 2 (Experimental): * Carboplatin-paclitaxel day1, q3 weeks, 6x, plus
  * Tumor Infiltrating Lymphocytes (TIL) starting 14 days after the 2nd chemotherapy cycle, q3 weeks, 3x, plus
  * Interferon Alpha 2A (3x10e6 U daily) starting one week before the first TIL infusion for 12 weeks in total.
  Interventions: Biological: Tumor Infiltrating Lymphocytes (TIL); Drug: Interferon Alfa 2A; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Biological: Tumor Infiltrating Lymphocytes (TIL) — Adoptive cell therapy using Tumor-Infiltrating Lymphocytes (TIL) i.v.
Drug: Interferon Alfa 2A — Interferon alpha (IFNα) s.c., may work as a low toxic preconditioning regimens that creates the space required for the infused TIL but that it also supports the TIL by sustaining their persistence and indirectly their function, by upregulation of HLA class I on tumor cells and decreasing the numbers of regulatory T cells.
  Other Names: IFNalpha
  Arms: Cohort 2
Drug: Carboplatin — chemotherapy i.v.
  Other Names: carboplatine
Drug: Paclitaxel — Chemotherapy i.v.
  Other Names: Taxol

SUMMARY:
The clinical benefit of standard treatment for patients with epithelial ovarian cancer (EOC) are poor. Ovarian cancer is a highly immunogenic tumor and good survival is tightly linked to the presence of tumor-infiltrating CD8+ T cells and the absence of immunosuppressive immune cells. This clear correlation between T cell infiltration and disease progression suggests that EOC may be sensitive to adoptive cell therapy by infusion of ex-vivo expanded autologous Tumor Infiltrating Lymphocytes (TIL) provided that immune suppression is reduced. Carboplatin+paclitaxel chemotherapy is directly killing tumor cells but was also shown to alleviate immunosuppression for 2 weeks coinciding with enhanced T-cell immunity, potentially creating a window of opportunity for T-cell based immunotherapy.

In addition, there is evidence that interferon alpha (IFNα) not only may work as a low toxic preconditioning regimens that creates the space required for the infused TIL but that it also supports the TIL by sustaining their persistence and indirectly their function, by upregulation of HLA class I on tumor cells and decreasing the numbers of regulatory T cells. Based on this we hypothesize that a synergistic clinical effect may be obtained when adoptive cell therapy with autologous TIL is administered during treatment with chemotherapy and IFNα. The feasibility and safety of TIL administration is studied in the window of opportunity created by carboplatin-paclitaxel chemotherapy with or without interferon alpha (IFNα). Furthermore, exploratory studies will be performed to analyze and confirm the proposed underlying mechanisms.

Tumor material for TIL production will be collected during first line debulking surgery in case of FIGO stage IIIC/IV disease (pre-OVACURE) or in case of recurrent platinum sensitive disease an extra biopsy can be planned (OVACURE).

DETAILED DESCRIPTION:
Study the feasibility and safety of TIL administration in the window of opportunity created by carboplatin-paclitaxel chemotherapy with or without interferon alpha (IFNα). Furthermore, exploratory studies will be performed to analyze and confirm the proposed underlying mechanisms.

Intervention:

Cohort 1

* Carboplatin-paclitaxel day1, q3 weeks, 6x, plus
* TIL starting 14 days after the 2nd chemotherapy cycle, q3 weeks, 3x.

Cohort 2

* Carboplatin-paclitaxel day1, q3 weeks, 6x, plus
* TIL starting 14 days after the 2nd chemotherapy cycle, q3 weeks, 3x, plus
* IFNα (3x10e6 U daily) starting one week before the first TIL infusion for 12 weeks in total.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Histologically proven epithelial ovarian cancer (EOC).
* Recurrent ovarian cancer amenable to carboplatin and paclitaxel chemotherapy. Patient with primary stage III or IV EOC can participate in the pre-OVACURE to collect rest tumor during debulking surgery for TILs preservation, so TILs will be available in case of recurrent disease will develop in the future.
* Presence of measurable progressive disease according to RECIST version 1.1 or elevated CA125 ≥ 2 times the upper normal limit (UNL) within 3 months and confirmed.
* Expected survival of at least 3 months.
* WHO performance status 0-2.
* Within the last 2 weeks prior to study day 0, vital laboratory parameters should be within normal range, except for the following laboratory parameters, which should be within the ranges specified:

Lab Parameter Range Hemoglobin ≥ 6,0 mmol/l Granulocytes ≥ 1,500/µl Lymphocytes ≥ 700/µl Platelets ≥ 100,000/µl Creatinine clearance ≥ 50 min/ml Serum bilirubin ≤ 40 mol/l ASAT and ALAT ≤ 5 times the normal upper limit LDH ≤ 2 times the normal upper limit

* Viral tests:

  * Negative for HIV type 1/2, HTLV and TPHA
  * No HBV (hepatitis B virus) antigen or antibodies against HBc in the serum
  * No antibodies against HCV (hepatitis C virus) in the serum
* Able and willing to give valid written informed consent.
* Prior treatment, including immunotherapy e.g. with anti-PD(L)1, is allowed but systemic therapy and radiotherapy must have been discontinued for at least two weeks before study entry.
* Patients should have disease progression.

Exclusion Criteria:

* Patients with brain metastases.
* Clinically significant heart disease (NYHA Class III or IV).
* Other serious acute or chronic illnesses, e.g. active infections requiring antibiotics, bleeding disorders, or other conditions requiring concurrent medications not allowed during this study.
* Active immunodeficiency disease or autoimmune disease requiring immune suppressive drugs. Vitiligo is not an exclusion criterion.
* Other malignancy within 2 years prior to entry into the study, except for treated non-melanoma skin cancer and in situ cervical or vulva carcinoma.
* Mental impairment that may compromise the ability to give informed consent and comply with the requirements of the study.
* Lack of availability for follow-up assessments.
* Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
NCI CTC criteria | 3 years
  If a DLT occurs in more than one out of the three patients, the study will be stopped. If < 1 out of 3 patients have a DLT, then three additional patients will be treated. Therefore, a minimum of 3 and a maximum of 6 patients will be treated in both cohorts.

SECONDARY OUTCOMES:
Clinical Response | 3 years
  Clinical response according to RECIST 1.1 criteria and immune response criteria (irRC)
Disease Control rate | 3 years
  Disease control rate (DCR: CR+PR+SD) at 6 months
Progression free survival (PFS) | 3 years
  Progression free survival (PFS) is defined as: the duration from the time of start chemotherapy until first observation of radiologically confirmed progressive disease or death due to any cause, whichever occurred first.
Overall Survival (OS) | 3 years
  Overall Survival (OS) is defined as: the duration from the time of start of chemotherapy until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Judith Kroep, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No